CLINICAL TRIAL: NCT03849300
Title: The Impacts of Aquatic Walking and Land-based Walking Exercise Therapy Programs on Vascular Function, Cardiorespiratory Capacity, Exercise Tolerance, Muscular Strength, and Physical Function in Patients With Peripheral Artery Disease
Brief Title: Impacts of Aquatic vs Land Walking on Vascular Health and Exercise Tolerance in Patients With Peripheral Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University (Other)
Collaborators: Marymount University (Other); Dong-Eui University (Other)
Responsible Party: Principal Investigator, Won-mok son, Principal Investigator, Pusan National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UNOmaha5
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Results first posted 2020-03-09 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Peripheral Artery Disease; Vascular Function; Exercise Tolerance; Peripheral Arterial Disease
Keywords: arterial stiffness; cardiorespiratory capacity; exercise tolerance; VO2max
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: aquatic walking exercise intervention group 1 vs. control group; aquatic walking exercise intervention group 2 vs. land-based walking exercise group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (No Intervention): No exercise intervention
- Aquatic walking exercise group 1 (Experimental): The aquatic walking exercise program was performed for 60 minutes per day, 4 times per week for 12 weeks.
  The program consisted of a warm-up (10 min) and cool-down (10 min) which included stretching and gait training. The 40-minute main exercise session included 10 minutes of hip flexion-extension, hip abduction-adduction, and knee flexion-extension. The last 30 minutes included water walking (forward, backward).
  The program intensity was established using heart rate reserve (HRR). Weeks 1-4 were at 50-60% HRR, weeks 5-8 were at 60-70% HRR, and weeks 9-12 were at 70-85% HRR. Subjects wore a heart rate monitor during the whole exercise training session in order to maintain the designated training intensity.
  Interventions: Other: Aquatic walking exercise program group 1
- Aquatic walking exercise group 2 (Experimental): The aquatic walking exercise program was performed for 60 minutes per day, 4 times per week for 12 weeks.
  The program consisted of a warm-up (10 min) and cool-down (10 min) which included stretching and gait training. The 40-minute main exercise session included 10 minutes of hip flexion-extension, hip abduction-adduction, and knee flexion-extension. The last 30 minutes included water walking (forward, backward).
  The program intensity was established using heart rate reserve (HRR). Weeks 1-4 were at 50-60% HRR, weeks 5-8 were at 60-70% HRR, and weeks 9-12 were at 70-85% HRR. Subjects wore a heart rate monitor during the whole exercise training session in order to maintain the designated training intensity.
  Interventions: Other: Aquatic walking exercise program group 2
- Land-based walking exercise group (Active Comparator): The land-based walking exercise program was performed for 60 minutes per day, 4 times per week for 12 weeks.
  The program consisted of a warm-up (10 min) and cool-down (10 min) which included stretching and gait training. The 40-minute main exercise session included 10 minutes of low-intensity forward, backward, and lateral side-stepping movements on flat group. The remaining 30 minutes included treadmill walking exercise.
  The program intensity was established using heart rate reserve (HRR). Weeks 1-4 were at 50-60% HRR, weeks 5-8 were at 60-70% HRR, and weeks 9-12 were at 70-85% HRR. Subjects wore a heart rate monitor during the whole exercise training session in order to maintain the designated training intensity.
  Interventions: Other: Land-based walking exercise group

INTERVENTIONS:
Other: Aquatic walking exercise program group 1 — 12 week aquatic walking exercise program
  Arms: Aquatic walking exercise group 1
Other: Aquatic walking exercise program group 2 — 12 week aquatic walking exercise program
  Arms: Aquatic walking exercise group 2
Other: Land-based walking exercise group — 12 week land-based walking exercise program
  Arms: Land-based walking exercise group

SUMMARY:
The purpose of this study was to examine the impacts of a 12-week aquatic walking exercise program on body composition, vascular function, cardiorespiratory capacity, exercise tolerance, muscular strength, and physical function in patients with peripheral artery disease (PAD). The effects of the 12-week aquatic walking exercise program were also compared to the effects of a 12-week land-based walking exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral artery disease (ankle-brachial index between 0.6 and 0.9)
* 50-85 years of age
* Sedentary (less than 1 hour of regular exercise participation per week within the previous year)

Exclusion Criteria:

* current smoker (smoking within previous 6 months)
* psychiatric conditions
* pulmonary disease
* renal disease
* thyroid disease

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2010-05-09 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2019-02-04 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Aquatic Walking Exercise Group 1; Aquatic Walking Exercise Group 2: The aquatic walking exercise program was performed for 60 minutes per day, 4 times per week for 12 weeks.
  The program consisted of a warm-up (10 min) and cool-down (10 min) which included stretching and gait training. The 40-minute main exercise session included 10 minutes of hip flexion-extension, hip abduction-adduction, and knee flexion-extension. The last 30 minutes included water walking exercise (forward, backward).
  The program intensity was established using heart rate reserve (HRR). Weeks 1-4 were at 50-60% HRR, weeks 5-8 were at 60-70% HRR, and weeks 9-12 were at 70-85% HRR. Subjects wore a heart rate monitor during the whole exercise training session in order to maintain the designated training intensity.
Period: Overall Study
Arm/Group | Control Group | Aquatic Walking Exercise Group 1 | Aquatic Walking Exercise Group 2 | Land-based Walking Exercise Group
Started | 42 | 42 | 32 | 31
Completed | 37 | 35 | 28 | 25
Not Completed | 5 | 7 | 4 | 6
Not completed — move out to different area | 1 | 3 | 1 | 4
Not completed — scheduling/transportation conflict | 4 | 4 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Land-based Walking Group: The land-based walking exercise program was performed for 60 minutes per day, 4 times per week for 12 weeks.
  The program consisted of a warm-up (10 min) and cool-down (10 min) which included stretching and gait training. The 40-minute main exercise session included 10 minutes of low-intensity forward, backward, and lateral side-stepping movements on flat group. The remaining 30 minutes included treadmill walking exercise.
  The program intensity was established using heart rate reserve (HRR). Weeks 1-4 were at 50-60% HRR, weeks 5-8 were at 60-70% HRR, and weeks 9-12 were at 70-85% HRR. Subjects wore a heart rate monitor during the whole exercise training session in order to maintain the designated training intensity.
- Total: Total of all reporting groups
Arm/Group | Control Group | Aquatic Walking Exercise Group 1 | Aquatic Walking Exercise Group 2 | Land-based Walking Group | Total
Number analyzed (Participants) | 42 | 42 | 32 | 31 | 147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 13 | 14 | 27
  >=65 years | 42 | 42 | 19 | 17 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (8) | 70 (10) | 70 (10) | 70 (10) | 70.1 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 42 | 32 | 31 | 147
  Male | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 42 | 42 | 32 | 31 | 147

OUTCOME MEASURES:

1. Primary Outcome: Peripheral Arterial Stiffness
Description: Peripheral arterial stiffness was estimated as measurement of femoral-to-ankle pulse wave velocity (meters per second). A higher value represents a worse outcome. Scale range is approximately 7.0 - 14.0 meters per second for healthy populations.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Control Group | Aquatic Walking Exercise Group 1 | Aquatic Walking Exercise Group 2 | Land-based Walking Exercise Group
Number analyzed (Participants) | 37 | 35 | 28 | 25
meters per second | 12.3 (1.1) | 10.2 (.9) | 12.4 (1.2) | 12.8 (1.4)

2. Secondary Outcome: Body Composition
Description: Body composition was measured using bioelectrical impedance analysis as percent body fat. A higher value represents a worse outcome. Scale range is approximately 10-35% for healthy populations.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: body fat percentage (%)
Arm/Group | Control Group | Aquatic Walking Exercise Group 1 | Aquatic Walking Exercise Group 2 | Land-based Walking Exercise Group
Number analyzed (Participants) | 37 | 35 | 28 | 25
body fat percentage (%) | 30.5 (5.2) | 28.5 (3.9) | 28.5 (5.2) | 28.7 (6.1)

3. Secondary Outcome: Resting Heart Rate
Description: Resting heart rate was measured as beats per minute (bpm). A higher value represents a worse outcome. Acceptable scale range is approximately 60-80 bpm for healthy populations.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Control Group | Aquatic Walking Exercise Group 1 | Aquatic Walking Exercise Group 2 | Land-based Walking Exercise Group
Number analyzed (Participants) | 37 | 35 | 28 | 25
beats per minute | 70.2 (10) | 67.9 (9) | 71 (5) | 71 (7)

4. Secondary Outcome: Systolic Blood Pressure
Description: Blood pressure was measured as millimeters of mercury (mmHg). Higher values represent a worse outcome. Scale range for systolic blood pressure is approximately 110-129mmHg for most healthy populations.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Control Group | Aquatic Walking Exercise Group 1 | Aquatic Walking Exercise Group 2 | Land-based Walking Exercise Group
Number analyzed (Participants) | 37 | 35 | 28 | 25
millimeters of mercury | 132.4 (9) | 130.4 (8.2) | 126 (9) | 129 (10)

5. Secondary Outcome: Resting Metabolic Rate
Description: Resting metabolic rate was measured as kilocalories per day. A higher value represents a better outcome. Scale range is approximately 1200-2200 kilocalories per day for healthy populations.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kilocalories per day
Arm/Group | Control Group | Aquatic Walking Exercise Group 1 | Aquatic Walking Exercise Group 2 | Land-based Walking Exercise Group
Number analyzed (Participants) | 37 | 35 | 28 | 25
kilocalories per day | 1022.9 (44.2) | 1021.5 (40.5) | 1282 (43) | 1272 (35)

6. Secondary Outcome: Cardiorespiratory Capacity
Description: Cardiorespiratory capacity was measured as the volume of maximal oxygen consumption in milliliters per kilogram per minute (VO2max, mL/kg/min). A higher value represents a better outcome. Scale range is approximately 25-60 mL/kg/min for healthy populations.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: milliliters/kilogram/minute of oxygen
Arm/Group | Control Group | Aquatic Walking Exercise Group 1
Number analyzed (Participants) | 37 | 35
milliliters/kilogram/minute of oxygen | 17.8 (5.3) | 20.5 (5.2)

7. Secondary Outcome: Exercise Tolerance - Walking Capacity
Description: Walking capacity was measured using the 6-minute walk test in meters. A higher value represents a better outcome. Scale range is approximately 400-1000 meters for healthy populations.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Control Group | Aquatic Walking Exercise Group 1 | Aquatic Walking Exercise Group 2 | Land-based Walking Exercise Group
Number analyzed (Participants) | 37 | 35 | 28 | 25
meters | 358 (92) | 440 (88) | 438 (97) | 404 (101)

8. Secondary Outcome: Upper Body Strength
Description: Upper body strength was measured as hand grip strength in kilograms (kg). A higher value represents a better outcome. Scale range is approximately 20-60kg for healthy populations.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Control Group | Aquatic Walking Exercise Group 1 | Aquatic Walking Exercise Group 2 | Land-based Walking Exercise Group
Number analyzed (Participants) | 37 | 35 | 28 | 25
kilograms | 25.1 (1.2) | 26 (3.7) | 26 (3) | 27 (5)

9. Secondary Outcome: Lower Body Strength
Description: Lower body strength was measured with leg extension in kilograms (kg). A higher value represents a better outcome. Scale range is approximately 20-120 kg for healthy populations.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Control Group | Aquatic Walking Exercise Group 1 | Aquatic Walking Exercise Group 2 | Land-based Walking Exercise Group
Number analyzed (Participants) | 37 | 35 | 28 | 25
kilograms | 45.2 (12.1) | 47.3 (20.9) | 48 (13) | 46 (11)

10. Secondary Outcome: Lower Body Flexibility
Description: Lower body flexibility was measured using sit-and-reach in centimeters (cm). A higher value represents a better outcome. Scale range is approximately 10-30 cm for healthy populations.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Control Group | Aquatic Walking Exercise Group 1
Number analyzed (Participants) | 37 | 35
centimeters | 15.2 (3.3) | 15.9 (6.3)

11. Secondary Outcome: Medical Outcomes Study Short-Form 36 General Health Survey for Physical Function
Description: The physical function domain score of the Medical Outcomes Study Short-Form 36 General Health Survey was measured. The scale range is from 0 to 100 percent. Higher scores represent a better outcome.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score in percents
Arm/Group | Control Group | Aquatic Walking Exercise Group 1 | Aquatic Walking Exercise Group 2 | Land-based Walking Exercise Group
Number analyzed (Participants) | 37 | 35 | 28 | 25
score in percents | 46 (21) | 52 (31) | 55 (27) | 53 (25)

12. Secondary Outcome: Diastolic Blood Pressure
Description: Blood pressure was measured as millimeters of mercury (mmHg). Higher values represent a worse outcome. Scale range for diastolic blood pressure is approximately 70-79 mmHg for most healthy populations.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Control Group | Aquatic Walking Exercise Group 1 | Aquatic Walking Exercise Group 2 | Land-based Walking Exercise Group
Number analyzed (Participants) | 37 | 35 | 28 | 25
millimeters of mercury | 90.7 (11) | 82.7 (10) | 84 (8) | 85 (10)

13. Secondary Outcome: Systemic Arterial Stiffness
Description: Systemic arterial stiffness was estimated as measurement of brachial-to-ankle pulse wave velocity (meters per second). A higher value represents a worse outcome. Scale range is approximately 7.0 - 14.0 meters per second for healthy populations.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: meters per second
Groups:
- Land-based Exercise Walking Group: The land-based walking exercise program was performed for 60 minutes per day, 4 times per week for 12 weeks.
  The program consisted of a warm-up (10 min) and cool-down (10 min) which included stretching and gait training. The 40-minute main exercise session included 10 minutes of low-intensity forward, backward, and lateral side-stepping movements on flat group. The remaining 30 minutes included treadmill walking exercise.
  The program intensity was established using heart rate reserve (HRR). Weeks 1-4 were at 50-60% HRR, weeks 5-8 were at 60-70% HRR, and weeks 9-12 were at 70-85% HRR. Subjects wore a heart rate monitor during the whole exercise training session in order to maintain the designated training intensity.
Arm/Group | Aquatic Walking Exercise Group 2 | Land-based Exercise Walking Group
Number analyzed (Participants) | 28 | 25
meters per second | 14.7 (1.9) | 14.8 (2.0)

14. Secondary Outcome: Time to Onset of Claudication
Description: Time to onset of claudication was measured during the 6-minute walking distance test (seconds). A higher value represents a better outcome. Healthy populations can typically walk the entire 6 minutes (360 seconds) without experiencing claudication.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Aquatic Walking Exercise Group 2 | Land-based Exercise Walking Group
Number analyzed (Participants) | 28 | 25
seconds | 252 (101) | 213 (99)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Control Group | Aquatic Walking Exercise Group 1 | Aquatic Walking Exercise Group 2 | Land-based Walking Group
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42 | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 0/32 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-05): https://cdn.clinicaltrials.gov/large-docs/00/NCT03849300/Prot_SAP_000.pdf